CLINICAL TRIAL: NCT05140694
Title: A Randomized, Active-comparator Controlled, Parallel-group Study, to Evaluate the Effect of Empagliflozin and Dulaglutide on MAFLD in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Empagliflozin and Dulaglutide on MAFLD in Patients With T2D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAFLD_empa_dula
Record Dates: First submitted 2021-04-26; First posted 2021-12-01 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Metabolic-associated Fatty Liver Disease; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; dulaglutide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Empagliflozin (Experimental): Empagliflozin 10mg p.o. once daily (available to control over ~25mg)
  Interventions: Drug: Empagliflozin
- Dulaglutide (Experimental): Dulaglutide 0.75mg s.c. once weekly (available to control over ~1.5mg)
  Interventions: Drug: Dulaglutide
- Empagliflozin and Dulagludie (Experimental): Empagliflozin 10mg p.o. once daily and dulaglutide 0.75mg s.c. once weekly
  Interventions: Drug: Empagliflozin and Dulaglutide

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10 mg p.o. once daily (available to control over ~25mg)
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Dulaglutide — Dulaglutide 0.75mg s.c. once a week (available to control over ~1.5mg)
  Other Names: Trulicity
  Arms: Dulaglutide
Drug: Empagliflozin and Dulaglutide — Empagliflozin 10 mg p.o. once daily with Dulaglutide 0.75mg s.c. once weekly
  Other Names: Jardiance and Trulicity
  Arms: Empagliflozin and Dulagludie

SUMMARY:
The co-administration of SGLT2 inhibitor and GLP-1 receptor agonist would be safe and effective on glycemic control in subjects with type 2 diabetes mellitus and MAFLD better than empagliflozin or dulaglutide alone.

The SGLT2 inhibitor and GLP-1 receptor agonist would be safe and effective on fatty liver disease in subjects with type 2 diabetes mellitus and MAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. age 20 or over
2. uncontrolled HbA1c (7~10%) with metformin and/or sulfonylurea
3. Hepatic steatosis estimated by Fibroscan (CAP ≥258 dB/m)
4. MAFLD: presence of any conditions

   1. Overweight or obese: BMI ≥23 kg/m2 (Asian)
   2. Metabolic dysregulation: at least of two of following criteria

      * Waist circumference: ≥90/80 cm in men and women (Asian)
      * Blood pressure ≥130/85 mmHg or drug treatment
      * Plasma triglycerides ≥150 mg/dL or drug treatment
      * Plasma HDL-cholesterol <40/50 mg/dL for men and women or drug treatment
      * Prediabetes (i.e. fasting glucose levels 100 to 125 mg/dL or 2-hour post-load glucose levels 140 to 199 mg/dL or HbA1c 5.7% to 6.4%
      * HOMA-insulin resistance score ≥2.5
      * Plasma high-sensitivity CRP >2 mg/L

Exclusion Criteria:

1. Significant alcohol consumption
2. Other competing causes for hepatic steatosis: viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha1 anti-trypsin deficiency, Celiac disease, Overt hypothyroidism, other secondary causes
3. Type 1 diabetes mellitus
4. medication usage within 3 months: vitamin E, PUFA, UDCA, fish oil, SGLT2 inhibitors, GLP1-RAs, TZDs
5. Severe organ dysfunction

   1. liver damage: AST/ALT >x5 UNL, albumin <3.2, platelet <60k, Child-Pugh-Turcotte stage B or C
   2. kidney damage: serum creatinine ≥2.0 mg/dL or eGFR <50 mL/min/1.72m2
6. Hepatocellular carcinoma, active tumor, or metastasis
7. End-stage liver disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of HbA1c level | baseline, week 12, week 24
  Patients achieving the target level
Changes of CAP score | baseline, week 24
  Controlled Attenuation Parameter (CAP) score by transient elastography

SECONDARY OUTCOMES:
Changes of LSM score | baseline, week 24
  Liver stiffness measurement (LSM) score by transient elastography
Changes of noninvasive liver fibrosis markers | baseline, week 12, week 24
  Noninvasive liver fibrosis markers will be calculated at baseline and at the end of the study
Changes of body weight and body composition | baseline, week 24
  Body composition by bioelectrical impedance will be measured at baseline and at the end of the study
Changes of lipid levels | baseline, week 12, week 24
  Cholesterol level will be measured at all visit days
Changes of ketone levels | baseline, week 12, week 24
  Ketone level will be measured at all visit days
Changes of liver parenchyma by ultrasonography | baseline, week 24
  improvement or deterioration
Changes of liver function parameters | baseline, week 12, week 24
  Liver enzymes, albumin will be measured at all visit days.
Changes of liver fibrosis biomarkers | baseline, week 24
  Type IV collagen
Changes of inflammation biomarker | baseline, week 24
  high-sensitivity CRP

OTHER OUTCOMES:
Changes of urine markers | baseline, week 12, week 24
  Urinalysis will be performed at all visit days
Changes of bone health | baseline, week 12, week 24
  parathyroid hormone, 25-hydroxylated vitamin will be measured at all visit days
Changes of gut microbiota | baseline, week 24
  gut microbiota composition, microbiota related to metabolic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital